CLINICAL TRIAL: NCT01603108
Title: Prospective Randomized Double Blind Placebo Controlled Trial of Rifaximin 550mg PO Twice Daily for Three Months to Prevent Recurrent Fibrosis in Liver Transplant Recipients With Chronic Hepatitis C Virus Infection
Brief Title: Rifaximin to Prevent Recurrent HCV-Related Fibrosis After Liver Transplant
Acronym: Rifaximin
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Elizabeth C. Verna, Assistant Professor of Medicine, Columbia University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: AAAI4155
Record Dates: First submitted 2012-04-26; First posted 2012-05-22 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: Hepatitis C
Keywords: Liver Transplant Recipient; Recurrent Fibrosis
MeSH Terms: conditions — Hepatitis C; Fibrosis | interventions — Rifaximin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rifaximin Arm (Experimental): Rifaximin will be initiated post-LT, once the subject is able to tolerate oral medications/diet. Rifaximin will be dosed at 550mg twice daily for 90 days (+/- 10 days) post-LT.
  Interventions: Drug: Rifaximin
- Placebo Control Arm (Placebo Comparator): Rifaximin placebo will be initiated post-LT, once the subject is able to tolerate oral medications/diet. Rifaximin placebo will be taken twice daily for 90 days (+/- 10 days) post-LT.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rifaximin — Rifaximin will be initiated post-LT, once the subject is able to tolerate oral medications/diet. Rifaximin will be dosed at 550mg twice daily for 90 days (+/- 10 days) post-LT.
  Other Names: Xifaxin
  Arms: Rifaximin Arm
Drug: Placebo — Rifaximin placebo will be initiated post LT, once the subject is able to tolerate oral medications/diet. Rifaximin placebo dosed at 550 mg twice daily for 90 days (+/10 days) post LT.
  Other Names: No other name
  Arms: Placebo Control Arm

SUMMARY:
The purpose of this study is to determine if the administration of a poorly-absorbable antibiotic (rifaximin) for the first three months after liver transplant will reduce the amount of fibrosis (or scarring of the liver) in liver transplant patients with recurrent hepatitis C virus (HCV) by lowering serum lipopolysaccharide (LPS), a protein in blood that comes from the bacteria in intestines and may cause scarring in the liver.

Approximately 60 subjects will participate in this study. Subjects will be part of the study for approximately 1 year post transplant.

DETAILED DESCRIPTION:
Hepatitis C virus (HCV) is the most common chronic liver infection and remains the leading indication for liver transplantation (LT). Although LT is a cure for cirrhosis of the liver, it does not always cure HCV infection or reinfection of post-transplanted liver. Post-LT recurrent HCV can lead to accelerated liver fibrosis. Chronic exposure to lipopolysaccharide (LPS) from gut-derived bacteria has shown to be at elevated levels in patients with cirrhosis due to HCV compared to normal controls. Therefore, the investigators hypothesize that LPS contributes to cause of liver fibrosis, specifically in patients with post-LT recurrent HCV, and this effect maybe modified with the poorly absorbed antibiotic, rifaximin, which alter the gut flora of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Subject must provide written informed consent before any study assessment is performed
* Age ≥ 18 years
* Willing and able to sign informed consent
* Chronic HCV infection with viremia
* Listed for liver transplantation
* Demonstrate ability to take oral medications prior to randomization (post LT)

Exclusion Criteria:

* Age < 18 years old
* Unwilling/able to sign informed consent
* Cleared HCV infection (and therefore not at risk for recurrent HCV)
* Human immunodeficiency virus (HIV) co-infection
* Hepatitis B (HBV) co-infection
* Participation in another interventional clinical trial
* Females of childbearing (reproductive) potential must have a negative serum pregnancy test at Screening and agree to use an acceptable method of contraception throughout their participation in the study
* Subjects with history of hypersensitivity to rifaximin, rifampin, rifamycin antimicrobial agents, or any of the components of rifaximin
* Subjects with history of tuberculosis infection or has received treatment for tuberculosis infection. If subject has previous positive test for tuberculosis antigen then they must have current negative chest x-ray to be eligible
* Subject has diarrhea and positive Clostridium difficile (C. difficile) toxin via stool examination during Screening period. NOTE: Stool examination for C. difficile toxin will be performed on subjects who have diarrhea during the screening period. Results of stool tests should be confirmed as negative prior to randomization

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2012-03; Primary Completion 2016-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Significant recurrence of Hepatitis C | One year post liver transplant
  Significant recurrence of hepatitis C at one year post-LT defined as at least stage 2 fibrosis, fibrosing cholestatic hepatitis or death/graft failure due to HCV.

SECONDARY OUTCOMES:
Measurement of Serum LPS | 3 months and 12 months post liver transplant
  Comparison of serum LPS measurements between groups, to determine if the use of rifaximin is associated with reduction in serum LPS.
Measurement of mRNA markers of the fibrosis cascade | 3 months and 12 months post liver transplant
  Comparison of mRNA markers of the fibrosis cascade between groups in the 3 month and 1 year post-LT liver biopsies.
Number of adverse events (severe and non-serious) | Up to 30 days post study participation
  Evaluation of the safety of Rifaximin compared to placebo in early post liver transplant patients, by assessing adverse events and severe adverse events experienced by the patients during the Rifaximin treatment course.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Verna, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center - NYPH, New York, New York, United States